CLINICAL TRIAL: NCT05415176
Title: Taurine Supplementation Associated or Not With Exercise: Effect on Browning of White Adipose Tissue in Elderly Women With Sarcopenic Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Taurine_exercise_browning
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Browning of Subcutaneous White Adipose Tissue Post Intervention; Metabolic and Inflammatory Variables Post Intervention
Keywords: Obesity; Sarcopenia; Brite adipose tissue; Taurine; Exercise
MeSH Terms: conditions — Obesity; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Taurine and Exercise (Tau+Exe) (Experimental): Individuals who will receive 3g of taurine supplementation combined with physical training in the period of 16 weeks
  Interventions: Dietary Supplement: Taurine supplementation; Other: Pshysical exercise
- Taurine (Tau) (Experimental): Individuals who will receive 3g of taurine supplementation
  Interventions: Dietary Supplement: Taurine supplementation
- Exercise (Exe) (Experimental): Individuals who will perform a physical training and receive a placebo supplementation in the period of 16 weeks
  Interventions: Other: Pshysical exercise
- Placebo (Cont) (Placebo Comparator): Individuals who will receive a placebo supplementation in the period of 16 weeks
  Interventions: Other: Placebo control

INTERVENTIONS:
Dietary Supplement: Taurine supplementation — Participants will receive 3g of taurine to be supplemented in the morning in single-dose capsules. The intervention will last 16 weeks.
  Arms: Taurine (Tau); Taurine and Exercise (Tau+Exe)
Other: Pshysical exercise — Participants will perform a multicomponent type workout that explores strength, aerobic and balance capacities with load progression every 15 days. The sessions will last 60 minutes each, being held three times a week with a day of rest in between. The intervention will last 16 weeks
  Arms: Exercise (Exe); Taurine and Exercise (Tau+Exe)
Other: Placebo control — The participants will receive a supplementation capsule containing placebo in the morning in single-dose capsules. The intervention will last 16 weeks.
  Arms: Placebo (Cont)

SUMMARY:
The aging process is followed by metabolic and body composition changes, increasing the risk of obesity and sarcopenia. The coexistence of these conditions acts synergistically on each other and is known as sarcopenic obesity. Beige adipose tissue is a tissue type that emerges from subcutaneous white adipose tissue (WAT), altering its phenotype to resemble the thermogenic functions of brown adipose tissue (BAT) in response to beta-adrenergic stimuli. Some in vitro and animal studies suggest that taurine supplementation and physical exercise are effective interventions in stimulating the aforementioned tissue, promoting what is known as WAT darkening, improving energy metabolism and showing benefits on the maintenance of muscle mass via stimulation of the coactivating protein PGC1α. These investigations are scarce in humans and could help health professionals in the adjuvant treatment of sarcopenic obesity. Therefore, the aim of the present study is to analyze the effects of taurine supplementation associated or not with physical exercise on the darkening of the WAT in sarcopenic obese elderly women.

DETAILED DESCRIPTION:
The aging process is followed by metabolic and body composition changes, increasing the risk of obesity and sarcopenia. The coexistence of these conditions acts synergistically on each other and is known as sarcopenic obesity. Beige adipose tissue is a tissue type that emerges from subcutaneous white adipose tissue (WAT), altering its phenotype to resemble the thermogenic functions of brown adipose tissue (BAT) in response to beta-adrenergic stimuli. Some in vitro and animal studies suggest that taurine supplementation and physical exercise are effective interventions in stimulating the aforementioned tissue, promoting what is known as WAT darkening, improving energy metabolism and showing benefits on the maintenance of muscle mass via stimulation of the coactivating protein PGC1α. These investigations are scarce in humans and could help health professionals in the adjuvant treatment of sarcopenic obesity. Therefore, the aim of the present study is to analyze the effects of taurine supplementation associated or not with physical exercise on the darkening of the WAT in sarcopenic obese elderly women. Volunteers with low appendicular lean mass (<15 kg) and body mass index (BMI) between 30 and 40 kg/m² will be recruited. These will be subdivided into 4 groups: control group (Cont), taurine (Tau), exercise (Exe) and exercise and taurine (Exe +Tau) and the duration of the intervention for all groups will be 16 weeks. Data related to anthropometry, body composition, biochemical tests, and food intake will be collected. To evaluate the effects on the darkening, a biopsy of the abdominal subcutaneous white adipose tissue will be performed to analyze protein, lipidomic and genetic parameters of this tissue pre and post intervention. Data will be analyzed by Analysis of Variance (ANOVA) or Kruskal-Wallis test depending on the normality of the data that will be tested by Shapiro-Wilk. A significance level for p <0.05 will be admitted. All analyzes will be performed in SPSS version 20 software.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 40kg/m²;
* Appendicular lean mass below 15 kg;
* Dynamometry below the cutoff point adjusted for sex and BMI (less than or equal to 21kg);
* "Sit and stand" test below the cut-off point adjusted for the age group, considering the number of repetitions in 30 seconds;
* Present medical certificate to perform physical exercise

Exclusion Criteria:

* alcoholics
* smokers
* diseases that prevents the practice of physical activity
* medical impediment to the practice of physical exercise throughout the study
* infectious diseases
* coronary diseases
* chronic kidney diseases
* undergoing nutritional monitoring or weight loss treatment
* score ≤13 for cognitive screening on the Mini-Mental State Examination (MMSE)

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 40 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Browning of white adipose tissue | 16 weeks
  Changes in the gene and protein expression on the subcutaneous white adipose tissue

SECONDARY OUTCOMES:
Changes in metabolic parameters - fasting blood glucose | 16 weeks
  Changes in fasting blood glucose samples in pre and post intervention
Changes in metabolic parameters - lipid profile | 16 weeks
  Changes in lipid profile (total cholesterol, HDL-c, LDL-c, triglycerides)samples in pre and post intervention
Changes in metabolic parameters - insulin sensitivity | 16 weeks
  Changes in insulin sensitivity samples in pre and post intervention
Body composition changes | 16 weeks
  Changes in fat-free mass and fat mass evaluated pre and post intervention by iDEXA
Improvement of physical performance | 16 weeks
  Improvement of physical performance evaluated by the 6-minute walk test, elbow flexion, sit and stand test and hand grip test
Indirect calorimetry assessment | 16 weeks
  Changes in resting metabolic rate (RMR) evaluated pre and post intervention by indirect calorimetry.
Changes in inflamatory markers | 16 weeks
  Evaluate the inflamatory markers PCR, IL-1β, IL-6, IL-10, IL-15, IFNy, MCP1, TNF-α, NFκβ, JNK1, PTP1B, iNOS
Changes in subcutaneous white adipose tissue (sWAT) morphology | 16 weeks
  Evaluate the changes in the white adipose tissue morphology by the histological analysis
Changes in Lipidomic profile of sWAT | 16 weeks
  Evaluate the fatty acids profile in the sWAT
Changes in plasma taurine | 16 weeks
  Evaluate the changes in the plasma taurine pre and post intervention
Changes in plasma irisin | 16 weeks
  Evaluate the changes in plasma irisin pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C de Freitas, PhD, Principal Investigator — University of São Paulo, School of Physical Education and Sports of Ribeirão Preto Ph.D. +55 16 3602-0345 ellenfreitas@usp.br
Locations (1):
- Escola de Educação Física e Esporte de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No